CLINICAL TRIAL: NCT05882383
Title: Changes of Optical Quality During the Peak of the Covid-19 Pandemic From November 2022 to January 2023 in China
Brief Title: Changes of Optical Quality During the Peak of the Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2023019
Record Dates: First submitted 2023-05-08; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Corneal Wavefront Aberration; SARS-CoV-2
Keywords: optical quality
MeSH Terms: conditions — Corneal Wavefront Aberration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: unifected with SARS-CoV-2 during follow-up
- Group A: uninfected at the first visit, have been infected at the second visit
- group B: have been infected at twice visit

SUMMARY:
To explore whether cornea structure, and optical quality are affected by the covid-19 infection.

DETAILED DESCRIPTION:
Participants with healthy corneas admitted to Tianjin Eye Hospital from November 25 to January 20, 2022 were followed up . At the end of the follow-up, the investigators recorded in detail whether the patients had undergone real-time reverse transcriptase polymerase chain reaction (covid-19 RT-PCR tests) testing, testing time and results. The presence of PCR-positive during follow-up is considered to be covid-19 infection; PCR-Negative and no symptoms of infection during the follow-up period are considered not infected; participants with symptoms but no PCR test were excluded from the study.Participants were divided into three groups according to the RT-PCR results and the presence or absence of symptoms of infection during follow-up. pentacam (Pentacam HR, Oculus, Wetzlar, Germany) was performed during follow-up and the results were recorded,and the data was statistically managed and compared.

ELIGIBILITY:
Included Criteria

1. Best corrected visual acuity (BCVA) ≥ 20/20;
2. No other eye diseases except myopia and astigmatism;
3. The cornea was transparent, and there was no cloud or pannus;
4. No clinical manifestation of Eye disease or systemic disease;

Exclusion Criteria:

1. corneal disease;
2. ocular trauma;
3. Pregnant and lactating women;

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients admitted to refractive center of Tianjin Eye Hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
The value of cornea aberration | 1 months
  The value of aberration data from pentacam during follow-up were compared, including coma, spherical aberration, defocus, and astigmatism
The value of cornea backscatter | 1 months
  The value of cornea backscatter from pentacam during follow-up were compared, including anterior layer，central layer and posterior
The value of cornea thickness | 1 months
  The value of cornea thickness from pentacam during follow-up were compared, includig the thinnest point, apex of the cornea.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Prof, Study Chair — Tianjin eye hosipital
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided